CLINICAL TRIAL: NCT05524389
Title: A Prospective Multicentre Phase III Randomised Open Clinical Study of Early Stage Endometrial Cancer Based on Molecular Classification and Traditional Risk Stratification to Guide Adjuvant Radiotherapy Decisions
Brief Title: Study of Early Stage Endometrial Cancer Based on Molecular Classification and Traditional Risk Stratification to Guide Adjuvant Radiotherapy Decisions
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: The First Affiliated Hospital of Air Force Medicial University (Other); The Second Affiliated Hospital of Dalian Medical University (Other); Second Hospital of Jilin University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); The Affiliated Hospital of Inner Mongolia Medical University (Other); Third Affiliated Hospital of Xinjiang Medical University (Other); Peking University First Hospital (Other); 940 Hospital of the People's Liberation Army Joint Logistic Support Force (Other); Xiangya Hospital of Central South University (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECMC-GART
Record Dates: First submitted 2022-08-30; First posted 2022-09-01 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-08

CONDITIONS: Endometrial Cancer; Adjuvant Radiotherapy; Molecular Classification
Keywords: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Observation; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Molecular classification based treatment (Experimental): Establishment of molecular-clinicopathological classification to make adjuvant treatment decisions: observation for favourable group; vaginal brachytherapy(VBT) for intermediate group; external beam radiotherapy(EBRT) for unfavourable group.
  Molecular-clinicopathological classification strategy：Favourable group：POLE-mutated. CTNNB1(wide-type)with IA (G1-3) or IB(G1-2)and LVSI(lymph-vascular space invasion) focal/-.
  Intermediate group：MMRD and LVSI focal/-. CTNNB1(wide-type) and IB(G3) or II with LVSI focal/-. CTNNB1-mutated and IA(G1-3) or IB (G1-2) with LVSI focal/-.
  Unfavourable group: TP53 mutation. CTNNB1-mutated and IB (G3) or II. Substantial LVSI.
  Interventions: Radiation: Vaginal brachytherapy; Radiation: Pelvic external beam radiotherapy; Other: Observation; Drug: Chemotherapy
- Conventional risk stratification based treatment (Active Comparator): Adjuvant vaginal brachytherapy alone for intermediate risk patients (IA G1-2 with LVSI present or age>60, IA G3 or IB G1-2 regardless of LVSI status).
  EBRT for high-intermediate risk (stage I B with G3, or stage II)
  Interventions: Radiation: Vaginal brachytherapy; Radiation: Pelvic external beam radiotherapy; Drug: Chemotherapy

INTERVENTIONS:
Radiation: Vaginal brachytherapy — High-dose rate vaginal brachytherapy (VBT) was delivered with a vaginal cylinder.For VBT administered alone, the dose is recommended: 3 fractions of 7 Gy or 5 fractions of 6 Gy or 6 fractions of 5 Gy.
  For VBT administered after completion of EBRT: 2-3 fractions of 4-6 Gy.
  Other Names: VBT
Radiation: Pelvic external beam radiotherapy — EBRT was delivered to the pelvic area using a total dose of 45-50.4Gy in 25-28 fractions over 5-6 weeks with the intensity-modulated radiotherapy (IMRT) technique, three-dimensional conformal radiotherapy (3D-CRT) modality
  Other Names: Pelvic EBRT
Other: Observation — No radiotherapy is administrated, but active follow-up and quality of life questionnaires is needed after surgery.
  Arms: Molecular classification based treatment
Drug: Chemotherapy — Intravenous concurrent or sequential adjuvant chemotherapy consists of carboplatin/paclitaxel, cisplatin/doxorubicin or cisplatin/doxorubicin/paclitaxel, etc.

SUMMARY:
The purpose of this study is to compare the efficacy and toxicity of early stage endometrial cancer based on molecular classification and conventional risk stratification adjuvant therapy decision-making, and to provide high-quality evidence-based medical evidence for individualized adjuvant therapy selection under the guidance of fine stratification system of endometrial cancer.

DETAILED DESCRIPTION:
This is an investigator-initiated prospective, national multicentre, phase III, randomised, open, non-inferiority clinical study. The study hypothesis is that adjuvant radiotherapy decision for early-stage endometrial cancer which is based on molecular classification can achieve de-escalation of adjuvant treatment without reducing local tumour control and survival, thereby potentially further reducing radiotherapy-related toxicity and improving quality of life, compared to using conventional risk stratification. The primary endpoint of this study is the 3-year local recurrence rate.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18-75.
2. Patients with newly histologically confirmed Endometrioid adenocarcinoma.
3. ECOG score 0-2
4. Surgery consisting of a total hysterectomy and bilateral salpingo-oophorectomy, pelvic lymphadenectomy or sentinel lymph node biopsy, with or without para-aortic lymphadenectomy, oophorectomy
5. Patients with FIGO staging(2009 edition) I or II and meet one of the following conditions:

   1. Stage IA G1-2 with massive LVSI+ or age ≥ 60 years
   2. Stage IA G3, regardless of LVSI status
   3. Stage IB G1-3, regardless of LVSI status
   4. Stage II, regardless of tumor grade and LVSI status
6. Patients can understand the study protocol and voluntarily participate in the study, and give written informed consent before treatment.

Exclusion Criteria:

1. Not FIGO stage I-II.
2. Residual tumor or positive margin.
3. Mixed carcinoma, sarcoma or carcinosarcoma
4. Previous history of malignant tumor
5. Previous history of pelvic radiotherapy
6. The interval between surgery and radiotherapy is more than 12 weeks.
7. With serious medical complications, such as heart disease, lung disease and other diseases that cannot tolerate the whole course of radiotherapy

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 624 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Loco-regional recurrence (LRR) | 3-year
  Loco-regional recurrence (LRR) is defined as the first recurrence in the vagina or pelvic cavity during follow-up, which was confirmed by imaging examination or biopsy pathology.

SECONDARY OUTCOMES:
Failure free survival(FFS) | 3-year,5-year
  FFS is defined as the time from randomization to recurrence,distant metastasis or death from any cause,whichever is first.
Overall survical(OS) | 3-year,5-year
  Overall survival is calculated from randomization to death from any cause.
Cumulative vaginal recurrence | 3-year,5-year
  Recurrence in the vaginal area during follow-up
Cumulative pelvic recurrence | 3-year,5-year
  Recurrence in the pelvic area, including the vagina, during follow-up
Distance metastasis(DM) | 3-year,5-year
  Distant metastasis (such as bone, lung, liver, brain, non-pelvic regional lymph node metastasis).
De-escalation rate of treatment | 3-year
  Comparison of the proportion of patients in two groups with the same clinicopathologic factors (FIGO, G, LVSI, age) downgraded from EBRT to VBT or from adjuvant radiotherapy (EBRT or VBT) to observation.
Health-related cancer-specific quality of life | 3-year,5-year
  General quality of life and general cancer related symptoms is accessed by Quality of Life Core Questionnaire (QLQC-30), ,scored as quite a bit/very much vs no or mild symptoms
Incidence of Acute and lateToxicities | 3-year,5-year
  Acute radiation enteritis, radiation cystitis, radiation lymphopenia, late radiation enteritis, radiation cystitis, vaginal stenosis or shortening, lymphedema, bone marrow suppression according to CTCAE v 5.0.
Endometrial cancer related health care costs | 3 years, 5 years
  All hospital based health care costs used with primary treatment or during follow-up for treatment of adverse events and/or treatment for relapse.

REFERENCES:
- [Background] Ren K, Wang W, Sun S, Hou X, Hu K, Zhang F. Recurrent patterns after postoperative radiotherapy for early stage endometrial cancer: A competing risk analysis model. Cancer Med. 2022 Jan;11(1):257-267. doi: 10.1002/cam4.4423. Epub 2021 Nov 15. PMID 34779587